CLINICAL TRIAL: NCT03812926
Title: Compuflo® Assisted Training vs Conventional Training for the Identification of the Ligamentum Flavum With an Epidural Simulator
Brief Title: Compuflo® vs Conventional Training With an Epidural Simulator
Status: Completed | Type: Observational
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Sponsor
Other Study IDs: EESOA1
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Epidural Simulator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Compuflo assited procedure — number of needle entry required to identify the ligamentum flavum
  Other Names: Standard assisted procedure

SUMMARY:
Epidural block is one of the most difficult skills that can be mastered by trainees probably due to the difficulty of recognizing the ligamentum flavum (LF) during the loss of resistance technique (LORT).The CompuFlo® Instrument can measure the pressure of human tissues in real-time at the orifice of a needle and it has been successfully used in clinical practice to identify the epidural space.The aim of this study was to evaluate whether Compuflo® may help trainees to identify the ligamentum flavum using a realistic Epidural Simulator

DETAILED DESCRIPTION:
The investigators enrolled 60 trainees who have never performed an epidural block. After having had a standardized learning module on epidural anatomy and technique, each trainee practiced the epidural and the Compuflo®-assisted LORT on the simulator for a maximum of 5 attemps. Trainees were asked to stop the needle entrance whenever they felt a sensation of an increase of resistance due to the penetration of the needle in the LF. The correct position of the needle was verified by an expert instructor. The number of attempts was noted. The power analysis required a sample size of 60 observations to set 80% test power and a 95% significance. Unpaired T-test was used to evaluate the differences in the number of epidural attempts. A logistic regression model was used to correlate the "success at the first attempt ratio" and the technique used.

ELIGIBILITY:
Inclusion Criteria:

First year trainees in anesthesia who never have performed an epidural block

Exclusion Criteria:

-

Ages: 26 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: First year trainees in anesthesia who never have performed an epidural block
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
epidural attempts | 10 minutes
  number of attempts to correctly identify the epidural space

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- EESOA Maternal Neonatal Simulation Centre, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capogna E, Coccoluto A, Gibiino G, Del Vecchio A. Compuflo(R)-Assisted Training vs Conventional Training for the Identification of the Ligamentum Flavum with an Epidural Simulator: A Brief Report. Anesthesiol Res Pract. 2019 Sep 12;2019:3804743. doi: 10.1155/2019/3804743. eCollection 2019. PMID 31611917